CLINICAL TRIAL: NCT02316275
Title: IMpact of Unrestricted ACTIVity Following Mid-Urethral Sling Surgery (I'M ACTIVe): Quality of Life and Cost Implications
Brief Title: Impact of Unrestrictive Exercise Following Mid-Urethral Sling Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer T. Anger, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00026474
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard post-operative activity restriction (Active Comparator): As a traditional method, patients will be restricted from activity for six weeks after sling surgery.
  Interventions: Other: Standard post-operative activity restriction
- No post-operative activity restrictions (Experimental): Patients are to resume regular activity immediately after mid-urethral sling surgery.
  Interventions: Other: No post-operative activity restrictions

INTERVENTIONS:
Other: No post-operative activity restrictions — Patients are to resume regular activity immediately after mid-urethral sling surgery. The investigators will determine the impact of unrestricted post-operative activity on continence outcomes of mid-urethral sling surgery in women with stress urinary incontinence (SUI). Investigators will measure the effect of unrestricted post-operative activity on early health-related quality of life (HRQOL). A Productivity Loss form for cost-effective analysis will be asked of the patient.
  Arms: No post-operative activity restrictions
Other: Standard post-operative activity restriction
  Arms: Standard post-operative activity restriction

SUMMARY:
To determine the impact of unrestricted postoperative activity on intermediate- and long-term continence outcomes of mid-urethral sling surgery in women with stress urinary incontinence.

To assess the natural return to baseline activity level when patients are unrestricted following mid-urethral sling surgery with or without concomitant anterior or posterior pelvic organ prolapse repair.

DETAILED DESCRIPTION:
Over the last decade, the mid-urethral sling has become the new gold standard in the management of stress urinary incontinence because of its high success rate and minimally invasive nature. However, postoperative management has not kept pace with the modernization of sling surgery. Although formal guidelines regarding the resumption of normal activity levels have not been established, it is general practice to restrict exercise for a minimum of six weeks after surgery.

For the study, if immediate resumption of normal activity has no impact on intermediate- and long-term continence outcomes, it may result in improved quality of life and cost savings from a societal perspective.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant female
* Self-reported stress urinary incontinence
* Incontinence demonstrated on physical exam and/or by an urodynamics study
* Planned mid-urethral sling surgery
* Available for 2 years of follow-up
* Willing and able to complete study assessments per the judgment of the treating clinician
* Willing and able to provide written informed consent

Exclusion Criteria:

* Age <18 years at time of enrollment
* Concomitant prolapse surgery other than anterior colporrhaphy
* Currently pregnant or <12 months post-partum
* Unable to read, write, or comprehend English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-12; Primary Completion 2021-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Unrestricted postoperative physical activity for surgical outcomes measure by questionnaire assessment. | 2 years
  Return to normal activity immediately after mid-urethral sling surgery could result in faster return to baseline health-related quality of life. Each questionnaire will be administered weekly following surgery until the patient returns to within 10% of baseline scores. Cost-effectiveness of early return to normal activity via Productivity Loss form as time spent recovering from surgery will be analyzed (incremental cost effectiveness ratio of net means by comparing the unrestricted and restricted groups).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Anger, MD, MPH, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Beverly Hills, California, United States

REFERENCES:
- [Background] Lose G, Jorgensen L, Thunedborg P. 24-hour home pad weighing test versus 1-hour ward test in the assessment of mild stress incontinence. Acta Obstet Gynecol Scand. 1989;68(3):211-5. doi: 10.3109/00016348909020991. PMID 2618603
- [Background] Herzog AR, Diokno AC, Brown MB, Normolle DP, Brock BM. Two-year incidence, remission, and change patterns of urinary incontinence in noninstitutionalized older adults. J Gerontol. 1990 Mar;45(2):M67-74. doi: 10.1093/geronj/45.2.m67. PMID 2313045
- [Background] Barber MD, Chen Z, Lukacz E, Markland A, Wai C, Brubaker L, Nygaard I, Weidner A, Janz NK, Spino C. Further validation of the short form versions of the Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ). Neurourol Urodyn. 2011 Apr;30(4):541-6. doi: 10.1002/nau.20934. Epub 2011 Feb 22. PMID 21344495
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Jenkinson C, Layte R, Jenkinson D, Lawrence K, Petersen S, Paice C, Stradling J. A shorter form health survey: can the SF-12 replicate results from the SF-36 in longitudinal studies? J Public Health Med. 1997 Jun;19(2):179-86. doi: 10.1093/oxfordjournals.pubmed.a024606. PMID 9243433
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Hynes DM, Stroupe KT, Luo P, Giobbie-Hurder A, Reda D, Kraft M, Itani K, Fitzgibbons R, Jonasson O, Neumayer L. Cost effectiveness of laparoscopic versus open mesh hernia operation: results of a Department of Veterans Affairs randomized clinical trial. J Am Coll Surg. 2006 Oct;203(4):447-57. doi: 10.1016/j.jamcollsurg.2006.05.019. Epub 2006 Jul 13. PMID 17000387
- [Background] Hamidi V, Andersen MH, Oyen O, Mathisen L, Fosse E, Kristiansen IS. Cost effectiveness of open versus laparoscopic living-donor nephrectomy. Transplantation. 2009 Mar 27;87(6):831-8. doi: 10.1097/TP.0b013e318199cfc9. PMID 19300185
- [Background] Laupacis A, Feeny D, Detsky AS, Tugwell PX. How attractive does a new technology have to be to warrant adoption and utilization? Tentative guidelines for using clinical and economic evaluations. CMAJ. 1992 Feb 15;146(4):473-81. PMID 1306034